CLINICAL TRIAL: NCT06598553
Title: What Works to Prevent Violence Against Women and Girls in Madagascar: Evaluation of Projet Jeune Leaders Comprehensive Sexual Education Curriculum in Rural Middle Schools
Brief Title: What Works to Prevent Violence Against Women and Girls in Madagascar
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Projet Jeune Leader (Unknown); United Kingdom Foreign Commonwealth Development Office (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00452498
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Comprehensive Sexual Education
Keywords: sexual education; adolescents; violence prevention; health

STUDY DESIGN:
Intervention Model Description: Hybrid effectiveness-implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Sexual Education (Experimental): All adolescents enrolled in intervention middle schools receive the 22 week program.
  Interventions: Behavioral: Projet Jeune Leader Comprehensive Sexual Education
- Usual educational program (No Intervention): Usual education program

INTERVENTIONS:
Behavioral: Projet Jeune Leader Comprehensive Sexual Education — PJL provides trained educators to deliver a 22 week comprehensive sexual education (CSE) curriculum in participating middle schools. All adolescents enrolled in the school receive the CSE program.
  Arms: Comprehensive Sexual Education

SUMMARY:
The study will evaluate a comprehensive sexual education program (CSE) delivered by Projet Jeune Leader (PJL), a women-led non-governmental program in Madagascar. The study will randomize 50 rural middle schools (grades 6-9), to either intervention (n=25) and control (n=25) schools. The CSE program will be implemented in the 25 intervention middle schools over the course of the school year (Sept-May) by trained PJL educators. Trained research assistants will conduct individual surveys at the beginning of the school year (baseline) and at the end of the school year (endline) with all students (ages 10-older) in both intervention and control schools. All student must have parental permission and provide informed consent to participate in the study, The surveys will include questions on demographics (e.g. age, sex/gender, grade, living situation), self-efficacy, bullying, physical abuse/violence, sexual harassment, sexual abuse and violence, harsh discipline at school and at home, gender/social norms, mental health and sexual and reproductive health. Teachers/school directors will also participate in the surveys, completing surveys at the beginning and end of the school year. The teacher/directors surveys will focus on health and safety of the students and school environment. In addition to the surveys, trained research assistants will conduct midline and endline qualitative interviews with a subsample of students, teachers and directors in the intervention schools to further explore the CSE intervention and impact on health and safety for students and teachers/directors.

DETAILED DESCRIPTION:
Projet Jeune Leader (PJL) - a southern-based, youth-founded, women-led, women's rights organization - has mainstreamed gender-transformative comprehensive sexuality education (CSE) in Madagascar's public schools. PJL's mission is to improve adolescent learning and well-being - especially in rural and under-served communities. Comprehensive sexuality education (CSE) plays an important role in transforming harmful gender norms and reducing the risk of violence. As an evidence- and curriculum-based intervention, CSE supports youth in developing knowledge, attitudes, skills, intentions, and behaviors for safe, healthy, and gender equitable relationships. PJL's CSE intervention, in particular, has been shown to improve young and very young adolescent students' knowledge, attitudes, self-efficacy, and behavioral intentions toward sexual and reproductive health and rights and gender equality using pre-post school year evidence with comparison schools (Projet Jeune Leader impact summary, 2024). Community-engaged participatory research using Human-centered design (HCD) tools has also revealed that the intervention is impacting aspects of human development which can underpin violence prevention and response, including but not limited to increasing students' courage and confidence, enhancing student-teacher relationships, strengthening family relationships, providing role models in the community, and facilitating the fight against drugs and violence in the community.

Through a formal partnership signed May 2022, Madagascar's National Ministry of Education has committed to institutionalize PJL's model into the education system to reach all schools, especially those that serve the 80% of Madagascar's population living in rural areas. PJL's multi-level partnership with Madagascar's Ministry of Education is unique, and PJL is well-positioned to implement action-oriented research to examine the effect of their CSE intervention on key outcomes of young adolescent victimization and/or perpetration of bullying and violence, and knowledge, attitudes and self-efficacy on violence, gender equality, strengths and difficulties (mental health) and sexual and reproductive health. PJL will also explore the CSE intervention's indirect effects on young adolescent school outcomes (retention, progression) and "safe school environment." Further, CSE implementation reach, implementation, adoption and maintenance with participating middle schools.

The evaluation of the PJL CSE intervention will be conducted through a collaboration between Johns Hopkins University and PJL.The study will use a hybrid type 2 effectiveness-implementation design guided by the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework. School-based surveys will be used to measure outcomes at baseline (beginning of school year) and endline (end of school year, 9 months post baseline) with adolescents in 6th-9th grades, teachers and directors at middle schools randomized to either intervention or control schools in targeted rural areas. In addition, quantitative and qualitative methods at midline and endline will be used to measure CSE intervention reach, adoption, implementation and maintenance in intervention middle schools.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 years or older
* Adolescents enrolled in grades 6th-9th in participating intervention and control middle schools in targeted districts
* Teachers and Directors in intervention and control middle schools in targeted districts
* Parent and adolescent provide Informed consent
* Teacher/director provides informed consent

Exclusion Criteria:

* Less than 10 years old
* Not a student intervention or control middle schools
* Not a teacher/director at intervention or control middle schools
* No informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Peer-to-peer violence victimization | Baseline, Post-baseline 9 months
  Score range 1-5; higher score indicates more experiences of peer to peer violence
Bullying | Baseline, Post-baseline 9 months
  Score range 1-5; higher score indicates more experiences of bullying
Dating violence | Baseline, Post-baseline 9 months
  Score range 1-5, higher score more experiences of dating violence
Harsh discipline in school | Baseline, Post-baseline 9 months
  Score range 1-5, higher score more experiences of harsh discipline

SECONDARY OUTCOMES:
Sexual health confidence | Baseline, Post-baseline 9 months
  Score range 1-4; higher score greater sexual health confidence
Gender equality | Baseline, Post-baseline 9 months
  Score range 1-4; higher score more gender equitable beliefs
Attitudes about dating violence/partner violence | Baseline, Post-baseline 9 months
  Score range 1-4; higher score indicates attitudes less endorsement of dating violence/partner violence
Self-confidence | Baseline, Post-baseline 9 months
  Score range 1-4; higher score greater self-confidence
Attitudes about healthy relationships | Baseline, Post-baseline 9 months
  Score range 1-4; higher score indicates attitudes that endorse healthy relationships
Mental Health (Strengths and Difficulties) | Baseline, Post-baseline 9 months
  Score range 1-3; higher score indicates better mental health

OTHER OUTCOMES:
Witness partner violence in home | Baseline, Post-baseline 9 months
  Score range 1-5; higher score indicates witness more intimate partner violence (IPV) at home
Parental Support | Baseline, Post-baseline 9 months
  Score range 1-4; higher score indicates greater parental support
Harsh discipline in home | Baseline, Post-baseline 9 months
  Score range 1-5; higher score indicates experiences of more harsh punishment in the home
Food security | Baseline, Post-baseline 9 months
  Score range 1-4; higher score indicates greater food insecurity

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Projet Jeune Leader, Fiananransoa, Madagascar

IPD SHARING:
Plan to Share IPD: No